CLINICAL TRIAL: NCT04317144
Title: Web-based Follow-up to Former ICU Patients
Acronym: WIVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WIVA001
Record Dates: First submitted 2020-01-16; First posted 2020-03-23 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Post Intensive Care Unit Syndrome
Keywords: intensive care units; survivors; web-based

STUDY DESIGN:
Intervention Model Description: Longitudinal observational study.
Who Masked: Investigator
Masking Description: Randomization is a in-hospital after consent done by the researcher/ICU-nurse. The participant receives group-specific information after randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based follow-up programme (Active Comparator): Participant randomized to the Web-based follow-up programme receive access to web-portal called www.1177.se
  Interventions: Behavioral: Web-based follow-up programme.
- No follow-up. (Active Comparator): Participants does not receive the web-based follow-up programme. e-questionnaires are sent out.
  Interventions: Behavioral: No follow-up

INTERVENTIONS:
Behavioral: Web-based follow-up programme. — Participants who are randomized to the intervention-group will have access to web-based follow-up for one year. The programme includes short films of equipment used in intensive care e.g. ventilator, suction-device. Continous renal replacement therapy , central vein catheter among other things. About 15 short films with icu-staff talking and show how the equipment works and alarm sounds. The intervention also includes lectures about how the ICU works and what problems a critically ill patient can suffer from post-icu. There is a built-in conversation tool in the programme that can be used both by the participant and the staff who works with the follow-up programme. Questionnaires is sent out 2,6 and 12 month post-icu. The questions include PTSD, Depression, QoL and physical activity. At the end of the study, participants are sent a questionnaire asking for their experience using the web-based follow up programme.
  Arms: Web-based follow-up programme
Behavioral: No follow-up — Participants randomized to "no follow-up" receive e-questionnaires 2, 6 and 12 months post-ICU care. The questions are the same as in web-based follow-up intervention group and include PTSD, Depression, QoL and physical activity.
  Arms: No follow-up.

SUMMARY:
This study evaluates if a web-based 1-year programme is a useful method for follow-up intensive care survivors with short ICU-stay. Half of the participants are randomized into receiving the web-based follow-up while the other half will receive no follow-up.

DETAILED DESCRIPTION:
It is not uncommon for Intensive care survivors to have persisting, psychiatric, cognitive and physical impairments long time after the critical illness occurred. Today, nurse-led follow-up is used but the main focus is on patients with a ICU-stay for at least three days. This study evaluates ICU-survivors with a maximum ICU-stay for 72 hours.

Participants are randomized to the web-based one year follow-up programme and no follow-up. Both group receive questionnaire 2, 6 and 12 month after the end of their intensive care stay.

The web-based follow-up programme includes, short lectures that describes the intensive care e.g. hallucinations, memory loss and delirium. The programme also include short films that shows the medical equipment and how and why it´s used. Regular contact with ICU-nurse to discuss any upcoming problems.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* Treated at the ICU under the time of the study.
* Have a Bank-id (which is needed to log in to the website.)

Exclusion Criteria:

* Institutionalized due to severe cognitive deficit.
* Does not communicate in the Swedish language.
* Patient is moved from other ICU to ICU where study is being held.
* Patient is sent to another ICU from ICU where study is being held.
* No home address.
* Patient decline to participate in study.
* Patient is receiving psychiatric specialist care post-icu e.g. high suicide risk.
* Patient is receiving ICU-treatment due to violence and is under on-going police-investigation.
* Palliative care.
* Patient receiving in-hospital care for more than 4 weeks in a row (except patient who is cared for in physical rehab-clinic at the hospital).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-07 (Estimated)

PRIMARY OUTCOMES:
Web-based follow up post-ICU impact on participants mental status concerning PTSD compared with no follow-up. | Questionnaire will be sent out at 2, 6 and 12 month post-ICU.
  Participant fill in questionnaire; Impact of event scale-revised (IES-R) which is screening for PTSD
Web-based follow up post-ICU impact on participants mental status regarding depression | Questionnaire will be sent out at 2, 6 and 12 month post-ICU.
  Patient Health Questionnaire (PHQ-9) which is screening for depression
Web-based follow up post-ICU impact on participants ability to deal with health related problems | Questionnaire will be sent out at 2, 6 and 12 month post-ICU.
  World Health Organization Disability Assessment Schedule (WHODAS 2.0) is a questionnaire which measure difficulties dealing with health-related problems.
Web-based follow-up post-ICU impact on participants physical activity level compared with no follow-up? | Questionnaires are sent out at 2, 6 and 12 month post-ICU.
  Participant answer one questionnaire; level of physical activity pre- and post ICU.
Participants will be asked what their opinions is on using web-based follow-up. | Questionnaire are sent at the end of the study-period.
  Semi-structured form

SECONDARY OUTCOMES:
Participants will be asked if they have unexpected hospital visit with health issues related to their ICU-stay. | This question is sent out at 2, 6 and 12 month post-ICU.
  Question sent out: Have you had unexpected hospital visits with health issues related to their ICU-stay.

CONTACTS AND LOCATIONS:
Overall Officials: Per Hellman, Phd, Study Chair — Uppsala University
Locations (1):
- Uppsala University hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olsson SJ, Ekblom O, Andersson E, Borjesson M, Kallings LV. Categorical answer modes provide superior validity to open answers when asking for level of physical activity: A cross-sectional study. Scand J Public Health. 2016 Feb;44(1):70-6. doi: 10.1177/1403494815602830. Epub 2015 Sep 21. PMID 26392418
- [Background] Vad är Intensivvård - SIR-Svenska Intensivvardsregistret [Internet]. [citerad 23 april 2018]. available at: http://www.icuregswe.org/sv/For-patienter/Vad-ar-Intensivvard/
- [Background] Pfoh ER, Wozniak AW, Colantuoni E, Dinglas VD, Mendez-Tellez PA, Shanholtz C, Ciesla ND, Pronovost PJ, Needham DM. Physical declines occurring after hospital discharge in ARDS survivors: a 5-year longitudinal study. Intensive Care Med. 2016 Oct;42(10):1557-1566. doi: 10.1007/s00134-016-4530-1. Epub 2016 Sep 16. PMID 27637716
- [Background] Hofhuis JG, Spronk PE, van Stel HF, Schrijvers AJ, Rommes JH, Bakker J. Experiences of critically ill patients in the ICU. Intensive Crit Care Nurs. 2008 Oct;24(5):300-13. doi: 10.1016/j.iccn.2008.03.004. Epub 2008 May 9. PMID 18472265
- [Background] Samuelson K, Lundberg D, Fridlund B. Memory in relation to depth of sedation in adult mechanically ventilated intensive care patients. Intensive Care Med. 2006 May;32(5):660-7. doi: 10.1007/s00134-006-0105-x. Epub 2006 Mar 7. PMID 16520999
- [Background] Svenningsen H, Egerod I, Dreyer P. Strange and scary memories of the intensive care unit: a qualitative, longitudinal study inspired by Ricoeur's interpretation theory. J Clin Nurs. 2016 Oct;25(19-20):2807-15. doi: 10.1111/jocn.13318. Epub 2016 Jul 26. PMID 27457029
- [Background] Myhren H, Ekeberg O, Toien K, Karlsson S, Stokland O. Posttraumatic stress, anxiety and depression symptoms in patients during the first year post intensive care unit discharge. Crit Care. 2010;14(1):R14. doi: 10.1186/cc8870. Epub 2010 Feb 8. PMID 20144193
- [Background] Peris A, Bonizzoli M, Iozzelli D, Migliaccio ML, Zagli G, Bacchereti A, Debolini M, Vannini E, Solaro M, Balzi I, Bendoni E, Bacchi I, Trevisan M, Giovannini V, Belloni L. Early intra-intensive care unit psychological intervention promotes recovery from post traumatic stress disorders, anxiety and depression symptoms in critically ill patients. Crit Care. 2011;15(1):R41. doi: 10.1186/cc10003. Epub 2011 Jan 27. PMID 21272307
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] de Azevedo JR, Montenegro WS, Rodrigues DP, de C Souza SC, Araujo VF, de Paula MP, Prazeres PH, da Luz Leitao A, Mendonca AV. Long-term cognitive outcomes among unselected ventilated and non-ventilated ICU patients. J Intensive Care. 2017 Feb 17;5:18. doi: 10.1186/s40560-017-0213-4. eCollection 2017. PMID 28239475
- [Background] Choi J, Hoffman LA, Schulz R, Tate JA, Donahoe MP, Ren D, Given BA, Sherwood PR. Self-reported physical symptoms in intensive care unit (ICU) survivors: pilot exploration over four months post-ICU discharge. J Pain Symptom Manage. 2014 Feb;47(2):257-70. doi: 10.1016/j.jpainsymman.2013.03.019. Epub 2013 Jul 12. PMID 23856099
- [Background] Ramnarain, D., Rutten, A., Van der Nat, G. et al. The impact of post intensive care syndrome in patients surviving the ICU: the downside of ICU treatment. ICMx 3, A530 (2015) doi:10.1186/2197-425X-3-S1-A530
- [Background] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703
- [Background] Sharshar T, Bastuji-Garin S, Stevens RD, Durand MC, Malissin I, Rodriguez P, Cerf C, Outin H, De Jonghe B; Groupe de Reflexion et d'Etude des Neuromyopathies En Reanimation. Presence and severity of intensive care unit-acquired paresis at time of awakening are associated with increased intensive care unit and hospital mortality. Crit Care Med. 2009 Dec;37(12):3047-53. doi: 10.1097/CCM.0b013e3181b027e9. PMID 19770751
- [Background] Wolters AE, Slooter AJ, van der Kooi AW, van Dijk D. Cognitive impairment after intensive care unit admission: a systematic review. Intensive Care Med. 2013 Mar;39(3):376-86. doi: 10.1007/s00134-012-2784-9. Epub 2013 Jan 18. PMID 23328935
- [Background] Schandl A, Bottai M, Holdar U, Hellgren E, Sackey P. Early prediction of new-onset physical disability after intensive care unit stay: a preliminary instrument. Crit Care. 2014 Jul 31;18(4):455. doi: 10.1186/s13054-014-0455-7. PMID 25079385
- [Background] Åkerman E, Fridh I, Orwelius L, Ringdal M, Shandl A. Nationella rekommendationer för uppföljning av patienter efter intensivvård. Riksföreningen Anestesi och intensivvård; 130617.
- [Background] Jensen JF, Thomsen T, Overgaard D, Bestle MH, Christensen D, Egerod I. Impact of follow-up consultations for ICU survivors on post-ICU syndrome: a systematic review and meta-analysis. Intensive Care Med. 2015 May;41(5):763-75. doi: 10.1007/s00134-015-3689-1. Epub 2015 Mar 3. PMID 25731633
- [Background] Glimelius Petersson C, Bergbom I, Brodersen K, Ringdal M. Patients' participation in and evaluation of a follow-up program following intensive care. Acta Anaesthesiol Scand. 2011 Aug;55(7):827-34. doi: 10.1111/j.1399-6576.2011.02474.x. Epub 2011 Jun 9. PMID 21658020
- [Background] Agard AS, Egerod I, Tonnesen E, Lomborg K. Struggling for independence: a grounded theory study on convalescence of ICU survivors 12 months post ICU discharge. Intensive Crit Care Nurs. 2012 Apr;28(2):105-13. doi: 10.1016/j.iccn.2012.01.008. Epub 2012 Feb 25. PMID 22365764
- [Background] Castillo MI, Cooke ML, Macfarlane B, Aitken LM. In ICU state anxiety is not associated with posttraumatic stress symptoms over six months after ICU discharge: A prospective study. Aust Crit Care. 2016 Aug;29(3):158-64. doi: 10.1016/j.aucc.2015.09.003. Epub 2015 Nov 6. PMID 26548628
- [Background] Hogberg KM, Sandman L, Nystrom M, Stockelberg D, Brostrom A. Caring Through Web-Based Communication: A Qualitative Evaluation of a Nursing Intervention to Create Holistic Well-Being Among Patients With Hematological Disease. J Holist Nurs. 2018 Sep;36(3):218-227. doi: 10.1177/0898010116667343. Epub 2016 Sep 22. PMID 27659277
- [Background] Wu RC, Delgado D, Costigan J, Maciver J, Ross H. Pilot study of an Internet patient-physician communication tool for heart failure disease management. J Med Internet Res. 2005 Mar 26;7(1):e8. doi: 10.2196/jmir.7.1.e8. PMID 15829480
- [Background] Stjernsward S, Hansson L. User value and usability of a web-based mindfulness intervention for families living with mental health problems. Health Soc Care Community. 2017 Mar;25(2):700-709. doi: 10.1111/hsc.12360. Epub 2016 May 17. PMID 27189237
- [Background] Sveen J, Low A, Dyster-Aas J, Ekselius L, Willebrand M, Gerdin B. Validation of a Swedish version of the Impact of Event Scale-Revised (IES-R) in patients with burns. J Anxiety Disord. 2010 Aug;24(6):618-22. doi: 10.1016/j.janxdis.2010.03.021. Epub 2010 Apr 12. PMID 20434306
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. The Patient Health Questionnaire Somatic, Anxiety, and Depressive Symptom Scales: a systematic review. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):345-59. doi: 10.1016/j.genhosppsych.2010.03.006. Epub 2010 May 7. PMID 20633738
- [Background] Carlozzi NE, Kratz AL, Downing NR, Goodnight S, Miner JA, Migliore N, Paulsen JS. Validity of the 12-item World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) in individuals with Huntington disease (HD). Qual Life Res. 2015 Aug;24(8):1963-71. doi: 10.1007/s11136-015-0930-x. Epub 2015 Jan 31. PMID 25636661
- [Background] Axelsson E, Lindsater E, Ljotsson B, Andersson E, Hedman-Lagerlof E. The 12-item Self-Report World Health Organization Disability Assessment Schedule (WHODAS) 2.0 Administered Via the Internet to Individuals With Anxiety and Stress Disorders: A Psychometric Investigation Based on Data From Two Clinical Trials. JMIR Ment Health. 2017 Dec 8;4(4):e58. doi: 10.2196/mental.7497. PMID 29222080